CLINICAL TRIAL: NCT02056171
Title: Efficacy of Quetiapine for Pediatric Delirium
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit subjects at our site within the past year.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1309014323
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Delirium
Keywords: delirium; pediatrics; critical care; quetiapine
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine (Experimental): A randomized group will receive quetiapine as treatment for delirium.
  Interventions: Drug: quetiapine
- Placebo (Placebo Comparator): A randomized group will receive placebo, and not quetiapine.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: quetiapine — Patients who are diagnosed with delirium and assigned to the intervention arm will receive quetiapine.
  Other Names: Seroquil
  Arms: Quetiapine
Other: Placebo — Patients who are diagnosed with delirium and assigned to the placebo arm will receive placebo.
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety and efficacy of quetiapine as treatment for pediatric delirium.

DETAILED DESCRIPTION:
Many children in the ICU become confused, due to their underlying illness or treatment effects. The medical term for this confusion is delirium. In adults, a medication called quetiapine has been effective in treating delirium. This is considered an "off label" use as the FDA has not approved quetiapine for this indication.

Pediatricians have been using quetiapine to treat delirium in children as well, but there is currently no data proving that it is effective in children. This study is being done to determine if quetiapine is effective for the treatment of ICU delirium in children.

ELIGIBILITY:
Inclusion Criteria:

- Any patient in the PICU aged 1 year to 21 years old who is diagnosed with delirium

Exclusion Criteria:

* Age <1
* Richmond Agitation Sedation Scale (RASS) score of -4 or -5 (deeply sedated or unarousable).
* current treatment for alcohol withdrawal
* hepatic encephalopathy
* pregnancy
* diagnosis of major depressive disorder or bipolar disorder
* diagnosis of movement disorder
* diagnosis of diabetic ketoacidosis
* baseline QTc >500 milliseconds
* non-English speaking subjects and/or parent/guardian

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chani Traube, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - NY Prebyterian Hospital/Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six participants were enrolled over 22 months between March 2015 and December 2016. The first participant was enrolled in March 2015 and the last participant was enrolled in December 2015.
Period: Overall Study
Arm/Group | Quetiapine | Placebo
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 18] | 3 [2 to 3] | 3 [2 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to First Resolution of Delirium
Description: Participants were screened for delirium daily. This describes the number of days from study drug initiation (either quetiapine or placebo) to first resolution of delirium (defined as a score of less than 9 on teh Cornell Assessment of Pediatric Delirium [CAPD]). If delirium did not resolve within the 10 day period, this defaults to 10 days.
Time Frame: Within the first 10 days after study enrollment
Population: All participants are included in analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 3 | 3
days | 8 [4 to 10] | 7 [2 to 10]

2. Secondary Outcome: Total ICU Days With Delirium
Description: Participants were screened for delirium daily. This describes the number of days with delirium within the 10 day study period.
Time Frame: Within 10 days after study enrollment
Measure: Mean (Full Range); unit: days
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 3 | 3
days | 8 [6 to 10] | 7 [2 to 10]

3. Other Pre Specified Outcome: Change in Delirium Severity
Description: Participants were screened for delirium daily using the Cornell Assessment for Pediatric Delirium, which assigns a delirium score between 0 (no delirium) to 32 (severe delirium). This describes the change in delirium score between study drug initiation (either quetiapine or placebo) and 72 hours. A decrease in score implies an improvement in delirium severity. For the quetiapine group, there was a median decrease in scale score (for the 3 subjects) of 1; for the placebo group, there was no change in delirium screen scores.
Time Frame: Baseline and 3 days of study drug initiation
Population: Change in CAPD score from baseline to day 3. A decrease in total score implies an improvement in delirium. An increase in total score implies worsening delirium.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 1 [1 to 2] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | Quetiapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=3) | Placebo (N=3)
movement disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No